CLINICAL TRIAL: NCT05522647
Title: Detection of Risk Behaviors: Pilot Observational Study With Bedridden and Agitated Patients.
Acronym: DECORIPAA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 DUBOIS; 2021-A03099-32 (Other: 2021-A03099-32)
Record Dates: First submitted 2022-08-18; First posted 2022-08-31 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Risk Behavior; Agitation; Hospitalization; Bedridden Patients
MeSH Terms: conditions — Risk-Taking; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
There is a risk of falls and injuries in bedridden hospitalized patients, increased in agitated or confused patients. In neurosurgery departments, brain damaged patients can present a loss of consciousness of risky behaviors and be in a state of agitation which frequently leads to their endangerment. The repercussions of this endangerment are multiple. For the patients, there may be a feeling of insecurity, with physical or chemical restraint solutions which deprive them of their freedom without a total guarantee of safety. For the caregivers, there is an emotional distress in front of this endangerment, and a professional guilt. Finally, there are economic repercussions due to the costs of complementary examinations and the lengthening of hospitalization.

The objective of the present study is to determine the nature and frequency of occurrence of risk behaviours, through the observation of bedridden and agitated hospitalized patients. These risk behaviours are defined as potentially dangerous and are warning signs for the caregiver. A better understanding of these behaviours could help to better anticipate falls and injuries and to implement preventive measures more quickly.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the Neurosurgery Department of the Clermont-Ferrand University Hospital
* Suffering from neurological and/or cognitive disorders leading to agitation and/or confusion
* Affiliation to a social security system
* Hospitalization in the department for at least 9 days
* Acceptance by the patient and/or trusted person capable of giving informed consent to participate in the research

Exclusion Criteria:

* Acute or transient agitation phase of somatic origin (bladder globe, pain, ionic disorder...)
* Patient under guardianship, curatorship or safeguard of justice
* Pregnant and breastfeeding women
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bedridden and agitated patients hospitalized in a neurosurgery department
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of risk behaviors observed per one-hour period | day 1
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 2
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 3
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 4
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 5
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 6
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 7
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 8
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.
Number of risk behaviors observed per one-hour period | day 9
  Each patient will be observed for 9 one-hour time slots, each distributed over a two-hour period between 6:00 am and midnight. The number of risk behaviors will be recorded for each one-hour observation period. Observation will be for one hour per day, with the order of the time slots randomly selected.

CONTACTS AND LOCATIONS:
Overall Officials: Charlène DUBOIS, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided